CLINICAL TRIAL: NCT04393597
Title: A Randomized, Open-label, Single-dose, Two-way Crossover Clinical Trial to Investigate the Effects of Food on the Pharmacokinetics of Orally Administered DWJ1458 in Healthy Adults
Brief Title: Effects of Food on the Pharmacokinetics of DWJ1458 in Healthy Adults
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: We decided to discontinue this particular clinical study through internal discussion.
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWJ1458102
Record Dates: First submitted 2020-05-13; First posted 2020-05-19 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Subjects take DWJ1458 on a fasted condition, and after wash-out period, take DWJ1458 with a high-fat diet.
  Interventions: Drug: DWJ1458 (fasted); Drug: DWJ1458 (fed)
- Group 2 (Experimental): Subjects take DWJ1458 with a high-fat diet, and after wash-out period, take DWJ1458 on a fasted condition.
  Interventions: Drug: DWJ1458 (fasted); Drug: DWJ1458 (fed)

INTERVENTIONS:
Drug: DWJ1458 (fasted) — Subjects take single dose of DWJ1458 on a fated condition
Drug: DWJ1458 (fed) — Subjects take single dose of DWJ1458 after high-fat diet

SUMMARY:
The purpose of this study is to evaluate the food effect on the pharmacokinetics of DWJ1458 after oral administration in healthy volunteers.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the food effect on the pharmacokinetics of DWJ1458 after oral administration in healthy volunteers: Randomized, open-label, oral, single-dose, crossover study

ELIGIBILITY:
Inclusion Criteria:

* Age 19 to 55 years
* BMI 18.5≥ and ≤27.0 kg/m²
* Female subjects must be menopause or surgically infertility.
* Male subjects must consent to contraception for at least 60 days after the study period and the final administration of the study drug.
* Those who understand the requirements of the study and sign a written informed consent, and also accept all the restrictions imposed during the course of the study.

Exclusion Criteria:

* History of hypersensitivity to investigational product
* Participation in a clinical drug study or bioequivalence study 6 months prior to the present study
* The subject who is judged to be unsuitable as a test subject in a screening test.
* The subject who is judged to be unsuitable for participation in a clinical trial due to other reasons determined by the investigators.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-28 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameter of DWJ1458: AUC0-t | 0 - 144 hours after dosing
  Area under the plasma concentration-time curve from time 0 to time t
Pharmacokinetic parameter of DWJ1458: Cmax | 0 - 144 hours after dosing
  Maximum plasma drug concentration

SECONDARY OUTCOMES:
Pharmacokinetic parameter of DWJ1458: AUCinf | 0 - 144 hours after dosing
  Area under the plasma concentration-time curve from drug administration to drug elimination
Pharmacokinetic parameter of DWJ1458: Tmax | 0 - 144 hours after dosing
  Time to reach maximum plasma concentration following drug administration
Pharmacokinetic parameter of DWJ1458: t1/2 | 0 - 144 hours after dosing
  Elimination half-life
Pharmacokinetic parameter of DWJ1458: Vd/F | 0 - 144 hours after dosing
  Apparent volume of distribution after oral administration
Pharmacokinetic parameter of DWJ1458: Cl/F | 0 - 144 hours after dosing
  Apparent total clearance of drug from plasma after oral administration

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No